CLINICAL TRIAL: NCT01932840
Title: Attitudes and Understanding of Plant Sterol Claims on Food Labels
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Advance Foods and Materials Network (Other)
Responsible Party: Principal Investigator, Mary R. L'Abbé, Earle W. McHenry Professor and Chair, Department of Nutritional Sciences, University of Toronto
Other Study IDs: AFMnet-01
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: General Population; Consumer Research
Keywords: attitudes and understanding of plant sterol claims; general Canadian population
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Canadian Consumer Monitor Panel: Canadian Consumer Monitor Panel is an online panel which answer surveys every 8-10 weeks about diet and health
  Interventions: Behavioral: Mock package questionnaire

INTERVENTIONS:
Behavioral: Mock package questionnaire — Within a online questionnaire we exposed participants randomly to 4 mock margarine packages differing only by the claim it carried and asked participants to answer several questions on attitudes and understanding after each mock package.

SUMMARY:
Daily consumption of plant sterols have been demonstrated to lower blood cholesterol. The Canadian government has recently allowed plant sterols to be added to certain foods and has also approved a disease risk reduction claim to be allowed on products containing plant sterols. However, it is unknown how Canadian consumers respond to plant sterol claims.

The objective of this study was to evaluate the attitudes and understanding of different types of plant sterol claims on food labels

ELIGIBILITY:
Inclusion Criteria:

* Primary grocery shoppers
* Canadian adults between the ages 20 to 69 years

Exclusion Criteria:

* Did not have an active email address or access to internet

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A subsection of the Canadian Consumer Monitor Panel - a national representative online consumer panel comprised of 30,000 Canadians
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response to survey questions measuring attitudes towards plant sterol claims using 5-point likert rating scales | On average the survey took 25 min to complete
  Within a online survey, participants were exposed to 4 mock margarine packages that differed only by the claim it carried. After being exposed to each mock package, participants were asked to rate their perceived attractiveness, healthiness, credibility, usefulness of the tested plant sterol claims using 5-point likert scales. Participants were also asked to rate their purchasing intentions of the mock margarine product with the different plant sterol claims.
Response to survey questions evaluating participants understanding of plant sterol claims | On average the survey took 25 minutes to complete
  After each mock package, understanding of plant sterol claims was evaluated using various survey methods. First, participants were asked to rate their perceived clarity of the wording of the claim using a 5-point likert scale (a subjective measure of understanding). Second, participants were ask to rate, on 5-point likert scales, the perceived benefit of consuming the mock margarine package for subgroups with different health conditions (an indirect measure of understanding). Finally we asked participants, in an open ended question, to explain what a claim means to a friend (an objective measure of understanding).

CONTACTS AND LOCATIONS:
Overall Officials: Mary R L'Abbé, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Guelph, Guelph, Ontario, Canada